CLINICAL TRIAL: NCT00205803
Title: A Phase I/II, 2-stage, Randomized, Double-Blind Trial of the Safety, Tolerability and Immunogenicity of 13-valent Pneumococcal Conjugate Vaccine (Serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) in Healthy Infants
Brief Title: Study Evaluating Pneumococcal Vaccine in Healthy Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6096A1-003
Record Dates: First submitted 2005-09-19; First posted 2005-09-20 (Estimated); Results first posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Subjects; Pneumococcal Infections
Keywords: Infant Vaccine
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

ARMS (2):
- 13vPnC (Experimental)
  Interventions: Biological: 13-Valent Pneumococcal Conjugate Vaccine (13vPnC)
- 7vPnC (Active Comparator)
  Interventions: Biological: 7-Valent Pneumococcal Conjugate Vaccine (7vPnC)

INTERVENTIONS:
Biological: 13-Valent Pneumococcal Conjugate Vaccine (13vPnC)
  Arms: 13vPnC
Biological: 7-Valent Pneumococcal Conjugate Vaccine (7vPnC)
  Arms: 7vPnC

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of the 13-valent pneumococcal conjugate vaccine (13vPnC) in healthy infants. This is the first study with this vaccine in infants.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6 weeks to 14 weeks (42-98 days of age) at time of enrollment,
2. In good health as determined by medical history, physical examination and judgment of the investigator,
3. Subject must have been born ≥36 weeks of gestational age,
4. Subject must be available for entire study period and whose parent/legal guardian can be reached by telephone,
5. Parent/legal guardian must be able to understand and sign an informed consent form prior to participation and complete a parent worksheet during study participation.

Exclusion Criteria:

1. Previous vaccination with licensed or investigational pneumococcal vaccine,
2. Previous vaccination with Hib conjugate, DTaP or IPV vaccines,
3. Contraindication to immunization with HepB, Hib conjugate, DTaP or IPV vaccines,
4. Significant neurological disorder or history of seizure including febrile seizure, or significant stable or evolving disorders such as cerebral palsy, encephalopathy, hydrocephalus or other significant disorders. Does not include resolving syndromes due to birth trauma such as Erb palsy,
5. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection,
6. History of culture-proven invasive disease caused by S. pneumoniae,
7. Previous anaphylactic reaction to any vaccine or vaccine components,
8. Major known congenital malformation or serious chronic disorders,
9. Participation in another investigational study (however, observation-only trials are permitted),
10. Known or suspected immune deficiency/suppression,
11. Receipt of blood products or gamma globulin (including Hepatitis B immunoglobulin and monoclonal antibody; eg, Synagis®).

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 249 (Actual)
Dates: Start 2004-09; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- New York, New York, United States

REFERENCES:
- [Derived] Bryant KA, Block SL, Baker SA, Gruber WC, Scott DA; PCV13 Infant Study Group. Safety and immunogenicity of a 13-valent pneumococcal conjugate vaccine. Pediatrics. 2010 May;125(5):866-75. doi: 10.1542/peds.2009-1405. PMID 20435707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the United States from September 2004 to September 2005.
Pre-assignment Details: Participants were enrolled into the study according to the inclusion/exclusion criteria without a screening period.
Groups:
- 13vPnC: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 2, 4, 6 months (infant series). Participants received one single 0.5mL dose of 13vPnC coadministered with ActHIB at 12-15 months of age (toddler dose).
- 7vPnC: Participants received one single 0.5mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with ActHIB and Pediarix at 2, 4, 6 months (infant series). Participants received one single 0.5mL dose of 7vPnC coadministered with ActHIB at 12-15 months of age (toddler dose).
Period: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 122 | 127
Vaccinated Dose 1 | 121 | 126
Vaccinated Dose 2 | 115 | 122
Vaccinated Dose 3 | 110 | 118
Completed | 104 | 116
Not Completed | 18 | 11
Not completed — Lost to Follow-up | 10 | 4
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Physician Decision | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost Kaiser coverage | 0 | 1
Not completed — Non-compliant | 1 | 0
Not completed — Sponsor request | 1 | 0
Period: After Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 104 | 116
Completed | 86 | 103
Not Completed | 18 | 13
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 3 | 2
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Other | 10 | 4
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 86 | 103
Completed | 84 | 100
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 121 | 126 | 247
Age Continuous [Mean (Standard Deviation); unit: weeks] | 9.2 (1.4) | 9.1 (1.2) | 9.2 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 117
  Male | 63 | 67 | 130

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions
Description: Local reaction events were collected using a paper worksheet. Tenderness was scaled as Any (tenderness present); Significant (Sig.) (present and interfered with limb movement). Induration and erythema were scaled as Any (induration or erythema present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (Mod.)(2.5 to 7.0 cm); Severe (Sev.)(> 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 15 days after each dose
Population: The safety population included all participants who received at least 1 dose of vaccine;(n)=number of participants with known values.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC Dose 1: Participants received one single 0.5mL dose of 13vPnC coadministered with Pediarix and ActHIB at 2 months of age (infant series Dose 1).
- 7vPnc Dose 1: Participants received one single 0.5mL dose of 7vPnC coadministered with Pediarix and ActHIB at 2 months of age (infant series Dose 1).
- 13vPnC Dose 2: Participants received one single 0.5mL dose of 13vPnC coadministered with Pediarix and ActHIB at 4 months of age (infant series Dose 2).
- 7vPnC Dose 2: Participants received one single 0.5mL dose of 7vPnC coadministered with Pediarix and ActHIB at 4 months of age (infant series Dose 2).
- 13vPnC Dose 3: Participants received one single 0.5mL dose of 13vPnC coadministered with Pediarix and ActHIB at 6 months of age (infant series Dose 3).
- 7vPnC Dose 3: Participants received one single 0.5mL dose of 7vPnC coadministered with Pediarix and ActHIB at 6 months of age (infant series Dose 3).
- 13vPnC Toddler Dose: Participants received one single 0.5mL dose of 13vPnC coadministered with ActHIB at 12 to 15 months of age (toddler dose).
- 7vPnC Toddler Dose: Participants received one single 0.5mL dose of 7vPnC coadministered with ActHIB at 12 to 15 months of age (toddler dose).
Arm/Group | 13vPnC Dose 1 | 7vPnc Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 121 | 126 | 115 | 122 | 110 | 118 | 86 | 103
percentage of participants
  Tenderness-Any (n=119,124,110,118,107,117,85,101) | 34.5 | 43.5 | 28.2 | 36.4 | 24.3 | 25.6 | 22.4 | 29.7
  Tenderness-Sig. (n=119,124,110,118,107,117,85,101) | 8.4 | 5.6 | 1.8 | 8.5 | 4.7 | 6.0 | 2.4 | 4.0
  Induration-Any (n=119,124,110,118,107,117,85,100) | 21.8 | 19.4 | 16.4 | 19.5 | 16.8 | 18.8 | 18.8 | 17.0
  Induration-Mild (n=119,123,110,117,107,116,85,100) | 20.2 | 17.9 | 16.4 | 17.1 | 16.8 | 17.2 | 18.8 | 17.0
  Induration-Mod. (n=119,123,110,117,107,116,85,100) | 3.4 | 2.4 | 3.6 | 3.4 | 0.0 | 4.3 | 2.4 | 3.0
  Induration-Sev. (n=119,123,110,117,107,116,85,100) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Erythema-Any (n=119,124,111,118,107,117, 85,100) | 21.0 | 19.4 | 16.2 | 17.8 | 17.8 | 19.7 | 24.7 | 19.0
  Erythema-Mild (n=119,124,110,117,106,116,85,99) | 20.2 | 19.4 | 13.6 | 17.1 | 16.0 | 18.1 | 24.7 | 16.2
  Erythema-Mod. (n=119,124,108,117,106,116,85,99) | 2.5 | 0.0 | 2.8 | 0.0 | 0.9 | 2.6 | 3.5 | 5.1
  Erythema-Severe (n=119,124,108,117,106,116,85,99) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

2. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events
Description: Systemic events (fever [Fv] ≥ 38 degrees Celsius [C] but ≤ 39 C, fever >39 C but ≤ 40 C, fever > 40 C, decreased (decr.) appetite, irritability, increased sleep, decreased sleep, use of medication (Med.)to prevent symptoms (sx), and use of medication to treat symptoms) were reported using a paper worksheet. Participants may be represented in more than 1 category.
Time Frame: Within 15 days after each dose
Population: The safety population included all participants who received at least 1 dose of vaccine; (n)=number of participants with known values.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Dose 1 | 7vPnc Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 121 | 126 | 115 | 122 | 110 | 118 | 86 | 103
percentage of participants
  Fv ≥38°C but≤39°C(n=114,121,102,114,100,113,78,94) | 16.7 | 16.5 | 21.6 | 24.6 | 20.0 | 20.4 | 14.1 | 12.8
  Fv >39°C but≤40°C(n=113,121,102,113,101,113,77,94) | 2.7 | 0.8 | 3.9 | 3.5 | 2.0 | 0.9 | 2.6 | 0.0
  Fv >40°C (n=113,121,102,113,100,113,76,94) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Decr. Appetite (n=118,124,110,118,107,117,85,101) | 30.5 | 31.5 | 22.7 | 22.9 | 27.1 | 30.8 | 22.4 | 21.8
  Decr. Sleep (n=118,124,110,118,107,117,84,101) | 18.6 | 17.7 | 24.5 | 19.5 | 21.5 | 18.8 | 13.1 | 14.9
  Increased Sleep (n=119,124,111,118,107,117,86,101) | 56.3 | 54.0 | 42.3 | 46.6 | 34.6 | 41.0 | 27.9 | 43.6
  Irritability (n=118,124,110,118,107,117,85,101) | 66.9 | 71.0 | 62.7 | 56.8 | 51.4 | 53.8 | 38.8 | 47.5
  Med.-Prevent Sx (n=95,101,86,96,83,93,85,102) | 29.5 | 33.7 | 34.9 | 32.3 | 36.1 | 43.0 | 17.6 | 35.3
  Med.-Treat Symptoms (n=94,101,86,96,84,94,85,101) | 44.7 | 34.7 | 48.8 | 50.0 | 42.9 | 47.9 | 29.4 | 27.7

3. Primary Outcome: Percentage of Participants Achieving Antibody Level ≥0.35μg/mL in 13vPnC Group Relative to 7vPnC Group After the 3-Dose Infant Series
Description: Percentage of participants achieving World Health Organization (WHO) predefined antibody threshold ≥0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: one month after 3-dose infant series (at 7 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n)=number of participants with a determinate postinfant series IgG antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 94 | 108
percentage of participants
  Common Serotypes - Serotype 4 (n=94,107) | 96.81 [90.96 to 99.34] | 99.07 [94.90 to 99.98]
  Common Serotypes - Serotype 6B (n=94,107) | 88.30 [80.03 to 94.01] | 88.79 [81.23 to 94.07]
  Common Serotypes - Serotype 9V (n=94,108) | 96.81 [90.96 to 99.34] | 99.07 [94.95 to 99.98]
  Common Serotypes - Serotype 14 (n=94,107) | 97.87 [92.52 to 99.74] | 97.20 [92.02 to 99.42]
  Common Serotypes - Serotype 18C (n=94,106) | 96.81 [90.96 to 99.34] | 99.06 [94.86 to 99.98]
  Common Serotypes - Serotype 19F (n=94,106) | 97.87 [92.52 to 99.74] | 97.17 [91.95 to 99.41]
  Common Serotypes - Serotype 23F (n=94,108) | 94.68 [88.02 to 98.25] | 95.37 [89.53 to 98.48]
  Additional Serotypes - Serotype 1 (n=94,108) | 97.87 [92.52 to 99.74] | 25.00 [17.17 to 34.25]
  Additional Serotypes - Serotype 3 (n=94,107) | 98.94 [94.21 to 99.97] | 14.02 [8.06 to 22.07]
  Additional Serotypes - Serotype 5 (n=93,107) | 100.00 [96.11 to 100.00] | 42.06 [32.58 to 51.99]
  Additional Serotypes - Serotype 6A (n=93,106) | 96.77 [90.86 to 99.33] | 33.96 [25.04 to 43.80]
  Additional Serotypes - Serotype 7F (n=94,105) | 98.94 [94.21 to 99.97] | 6.67 [2.72 to 13.25]
  Additional Serotypes - Serotype 19A (n=94,107) | 100.00 [96.15 to 100.00] | 94.39 [88.19 to 97.91]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For serotype 4 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = -2.26, 95% CI 2-sided [-8.08 to 2.33]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For serotype 6B the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = -0.49, 95% CI 2-sided [-9.93 to 8.65]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For serotype 9V the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = -2.27, 95% CI 2-sided [-8.07 to 2.26]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For serotype 14 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 0.68, 95% CI [-4.96 to 6.16]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For serotype 18C the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = -2.25, 95% CI [-8.18 to 2.36]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For serotype 19F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 0.70, 95% CI [-4.84 to 6.32]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For serotype 23F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = -0.69, 95% CI [-7.75 to 5.86]
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; For serotype 1 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 72.87, 95% CI [63.32 to 81.07]
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; For serotype 3 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 84.92, 95% CI [76.73 to 91.05]
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; For serotype 5 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 57.94, 95% CI [48.01 to 67.42]
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; For serotype 6A the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 62.81, 95% CI [52.33 to 72.20]
Statistical Analysis 12: Comparison: 13vPnC vs 7vPnC; For serotype 7F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 92.27, 95% CI [85.26 to 96.54]
Statistical Analysis 13: Comparison: 13vPnC vs 7vPnC; For serotype 19A the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 5.61, 95% CI [1.23 to 11.86]

4. Secondary Outcome: Percentage of Participants Achieving Antibody Level ≥0.35μg/mL in 13vPnC Group Relative to 7vPnC Group After the Toddler Dose
Description: Percentages of participants achieving WHO predefined antibody threshold ≥0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: One month after the toddler dose (at 13 to 16 months of age)
Population: The All-Available Toddler Immunogenicity population consisted of eligible participants who had at least 1 valid and determinate assay result related to the proposed analysis; (n)=number of participants with a determinate posttoddler dose IgG antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 85 | 102
percentage of participants
  Common Serotypes - Serotype 4 (n=78,94) | 97.4 [91.0 to 99.7] | 98.9 [94.2 to 100.0]
  Common Serotypes - Serotype 6B (n=78,93) | 100.0 [95.4 to 100.0] | 100.0 [96.1 to 100.0]
  Common Serotypes - Serotype 9V (n=78,94) | 98.7 [93.1 to 100.0] | 100.0 [96.2 to 100.0]
  Common Serotypes - Serotype 14 (n=78,93) | 100.0 [95.4 to 100.0] | 100.0 [96.1 to 100.0]
  Common Serotypes - Serotype 18C (n=78,94) | 100.0 [95.4 to 100.0] | 100.0 [96.2 to 100.0]
  Common Serotypes - Serotype 19F (n=78,93) | 100.0 [95.4 to 100.0] | 100.0 [96.1 to 100.0]
  Common Serotypes - Serotype 23F (n=78,93) | 100.0 [95.4 to 100.0] | 97.8 [92.4 to 99.7]
  Additional Serotypes - Serotype 1 (n=78,91) | 100.00 [95.4 to 100.00] | 2.2 [0.3 to 7.7]
  Additional Serotypes - Serotype 3 (n=78,92) | 92.3 [84.0 to 97.1] | 8.7 [3.8 to 16.4]
  Additional Serotypes - Serotype 5 (n=78,78) | 100.0 [95.4 to 100.0] | 70.5 [59.1 to 80.3]
  Additional Serotypes - Serotype 6A (n=78,92) | 100.0 [95.4 to 100.0] | 88.0 [79.6 to 93.9]
  Additional Serotypes - Serotype 7F (n=78,85) | 100.0 [95.4 to 100.0] | 5.9 [1.9 to 13.2]
  Additional Serotypes - Serotype 19A (n=78,93) | 100.0 [95.4 to 100.0] | 100.0 [96.1 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For serotype 4 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = -1.5, 95% CI [-7.9 to 3.6]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For serotype 6B the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 0.0, 95% CI [-4.6 to 4.0]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For serotype 9V the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = -1.3, 95% CI [-6.9 to 2.8]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For serotype 14 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 0.0, 95% CI [-4.6 to 4.0]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For serotype 18C the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 0.0, 95% CI [-4.7 to 3.9]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For serotype 19F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 0.0, 95% CI [-4.6 to 4.0]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For serotype 23F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 2.2, 95% CI [-2.6 to 7.7]
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; For serotype 1 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 97.8, 95% CI [92.3 to 99.7]
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; For serotype 3 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 83.6, 95% CI [73.2 to 90.8]
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; For serotype 5 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 29.5, 95% CI [19.7 to 40.9]
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; For serotype 6A the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 12.0, 95% CI [5.9 to 20.4]
Statistical Analysis 12: Comparison: 13vPnC vs 7vPnC; For serotype 7F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 94.1, 95% CI [86.8 to 98.1]
Statistical Analysis 13: Comparison: 13vPnC vs 7vPnC; For serotype 19A the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 0.0, 95% CI [-4.6 to 4.0]

5. Secondary Outcome: Geometric Mean Antibody Concentration in 13vPnC Group Relative to 7vPnC Group After the 3-Dose Infant Series
Description: Antibody geometric mean concentration (GMC) as measured by enzyme-linked immunosorbent assay (ELISA) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC ratios (13vPnC/7vPnC) and corresponding 2-sided 95% CI were evaluated.
Time Frame: One month after 3-dose infant series (at 7 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations;(n)=number of participants with a determinate antibody concentration for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 94 | 108
μg/mL
  Common Serotypes - Serotype 4 (n=94,107) | 1.81 [1.54 to 2.13] | 2.40 [2.01 to 2.87]
  Common Serotypes - Serotype 6B (n=94,107) | 2.74 [2.02 to 3.71] | 2.86 [2.09 to 3.91]
  Common Serotypes - Serotype 9V (n=94,108) | 1.52 [1.29 to 1.78] | 1.78 [1.55 to 2.05]
  Common Serotypes - Serotype 14 (n=94,107) | 4.24 [3.44 to 5.23] | 5.19 [4.13 to 6.52]
  Common Serotypes - Serotype 18C (n=94,106) | 1.53 [1.30 to 1.80] | 2.46 [2.08 to 2.91]
  Common Serotypes - Serotype 19F (n=94,106) | 2.21 [1.87 to 2.61] | 2.58 [2.17 to 3.08]
  Common Serotypes - Serotype 23F (n=94,108) | 1.39 [1.15 to 1.67] | 1.81 [1.51 to 2.19]
  Additional Serotypes - Serotype 1 (n=94,108) | 2.57 [2.14 to 3.08] | 0.06 [0.05 to 0.09]
  Additional Serotypes - Serotype 3 (n=94,107) | 1.40 [1.20 to 1.62] | 0.09 [0.07 to 0.11]
  Additional Serotypes - Serotype 5 (n=93,107) | 2.41 [2.07 to 2.80] | 0.28 [0.22 to 0.34]
  Additional Serotypes - Serotype 6A (n=93,106) | 2.36 [1.89 to 2.94] | 0.25 [0.20 to 0.30]
  Additional Serotypes - Serotype 7F (n=94,105) | 1.85 [1.62 to 2.11] | 0.07 [0.06 to 0.08]
  Additional Serotypes - Serotype 19A (n=94,107) | 1.93 [1.64 to 2.27] | 1.12 [0.96 to 1.32]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For serotype 4 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 0.76, 95% CI [0.59 to 0.96]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For serotype 6B the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 0.96, 95% CI [0.62 to 1.48]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For serotype 9V the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Difference = 0.85, 95% CI [0.69 to 1.05]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For serotype 14 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 0.82, 95% CI [0.60 to 1.11]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For serotype 18C the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 0.62, 95% CI [0.49 to 0.79]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For serotype 19F the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 0.86, 95% CI [0.67 to 1.09]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For serotype 23F the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 0.77, 95% CI [0.59 to 1.00]
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; For serotype 1 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 39.78, 95% CI [27.47 to 57.63]
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; For serotype 3 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 15.56, 95% CI [11.63 to 20.81]
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; For serotype 5 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 8.67, 95% CI [6.65 to 11.29]
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; For serotype 6A the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 9.60, 95% CI [7.07 to 13.04]
Statistical Analysis 12: Comparison: 13vPnC vs 7vPnC; For serotype 7F the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 26.78, 95% CI [20.97 to 34.22]
Statistical Analysis 13: Comparison: 13vPnC vs 7vPnC; For serotype 19A the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 1.71, 95% CI [1.36 to 2.16]

6. Secondary Outcome: Geometric Mean Concentration in 13vPnC Group Relative to 7vPnC Group Before and After the Toddler Dose
Description: Antibody geometric mean concentration (GMC) as measured by ELISA with their corresponding 95% CI immediately before and after the toddler dose for 7 common pneumococcal serotypes (Serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: Immediately before (12 to 15 months of age) and one month after the toddler dose (13 to 16 months of age)
Population: All-Available Toddler Immunogenicity population consisted of eligible participants who had at least 1 valid and determinate assay result related to proposed analysis;(n)= number of participants with a determinate antibody concentration for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- 13vPnC Before Toddler Dose: Participants received one single 0.5mL dose of 13vPnC coadministered with ActHIB and Pediarix at 2, 4, 6 months (infant series).
- 7vPnC Before Toddler Dose: Participants received one single 0.5mL dose of 7vPnC coadministered with ActHIB and Pediarix at 2, 4, 6 months (infant series).
- 13vPnC After Toddler Dose: Participants received one single 0.5mL dose of 13vPnC coadministered with ActHIB at 12-15 months of age (toddler dose).
- 7vPnC After Toddler Dose: Participants received one single 0.5mL dose of 7vPnC coadministered with ActHIB at 12-15 months of age (toddler dose).
Arm/Group | 13vPnC Before Toddler Dose | 7vPnC Before Toddler Dose | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 85 | 102 | 85 | 102
μg/mL
  Common Serotypes-Serotype 4 (n=83,100,78,94) | 0.33 [0.28 to 0.40] | 0.48 [0.41 to 0.56] | 2.86 [2.31 to 3.55] | 4.09 [3.34 to 5.00]
  Common Serotypes-Serotype 6B (n=82,98,78,93) | 0.84 [0.69 to 1.03] | 0.95 [0.77 to 1.18] | 11.03 [8.78 to 13.86] | 11.85 [9.63 to 14.56]
  Common Serotypes-Serotype 9V (n=83,100,78,94) | 0.43 [0.37 to 0.51] | 0.43 [0.37 to 0.50] | 2.55 [2.15 to 3.02] | 2.75 [2.37 to 3.18]
  Common Serotypes-Serotype 14 (n=83,100,78,93) | 1.59 [1.27 to 2.00] | 2.00 [1.66 to 2.41] | 7.68 [6.08 to 9.70] | 10.24 [8.23 to 12.74]
  Common Serotypes-Serotype 18C (n=83,100,78,94) | 0.25 [0.22 to 0.30] | 0.40 [0.34 to 0.46] | 2.57 [2.08 to 3.18] | 4.08 [3.42 to 4.87]
  Common Serotypes-Serotype 19F (n=82,100,78,93) | 0.81 [0.66 to 1.00] | 0.60 [0.49 to 0.72] | 6.34 [5.06 to 7.94] | 3.97 [3.26 to 4.85]
  Common Serotypes-Serotype 23F (n=83,100,78,93) | 0.29 [0.24 to 0.36] | 0.38 [0.31 to 0.47] | 3.36 [2.70 to 4.18] | 4.79 [3.86 to 5.94]
  Additional Serotypes-Serotype 1 (n=83,90,78,91) | 0.68 [0.56 to 0.82] | 0.04 [0.03 to 0.04] | 3.44 [2.79 to 4.23] | 0.03 [0.03 to 0.04]
  Additional Serotypes-Serotype 3 (n=83,98,78,92) | 0.27 [0.23 to 0.32] | 0.09 [0.07 to 0.12] | 1.11 [0.94 to 1.33] | 0.10 [0.08 to 0.12]
  Additional Serotypes-Serotype 5 (n=83,92,78,78) | 1.01 [0.87 to 1.18] | 0.40 [0.31 to 0.50] | 3.92 [3.27 to 4.69] | 0.56 [0.45 to 0.70]
  Additional Serotypes-Serotype 6A (n=82,96,78,92) | 0.81 [0.68 to 0.96] | 0.27 [0.22 to 0.33] | 8.06 [6.60 to 9.85] | 1.68 [1.27 to 2.21]
  Additional Serotypes-Serotype 7F (n=83,91,78,85) | 0.58 [0.50 to 0.67] | 0.04 [0.03 to 0.05] | 2.67 [2.26 to 3.16] | 0.05 [0.04 to 0.06]
  Additional Serotypes-Serotype19A (n=83,100,78,93) | 0.85 [0.67 to 1.09] | 0.64 [0.52 to 0.79] | 5.60 [4.60 to 6.83] | 2.82 [2.32 to 3.41]

7. Secondary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Haemophilus Influenzae Type b, Diphtheria Toxoid, Polio, Pertussis, Tetanus, and Hepatitis B in 13vPnC Group Relative to 7vPnC Group After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold levels for Haemophilus Influenzae Type b (Hib) polyribosylribitol phosphate (PRP), Diphtheria Toxoid, Polio (Types 1, 2, and 3), Pertussis (filamentous hemagglutinin [FHA], Pertussis Toxoid, and Pertactin), Tetanus, and Hepatitis B with the corresponding 95% CI for each concomitant antigen are presented.
Time Frame: One month after the infant series (7 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations;(n)=number of participants with a determinate postinfant series antibody level to the given concomitant vaccine component.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 94 | 108
Percentage of participants
  Hib (PRP) 0.15 μg/mL (n=84,87) | 89.29 [80.63 to 94.98] | 86.21 [77.15 to 92.66]
  Hib (PRP) 1.0 μg/mL (n=84,87) | 70.24 [59.27 to 79.73] | 63.22 [52.20 to 73.31]
  Diphtheria 0.01 IU/mL (n=38,48) | 100.00 [90.75 to 100.00] | 100.00 [92.60 to 100.00]
  Diphtheria 0.1 IU/mL (n=38,48) | 100.00 [90.75 to 100.00] | 100.00 [92.60 to 100.00]
  Tetanus 0.01 IU/mL (n=38,48) | 100.00 [90.75 to 100.00] | 100.00 [92.60 to 100.00]
  Tetanus 0.1 IU/mL (n=38,48) | 100.00 [90.75 to 100.00] | 100.00 [92.60 to 100.00]
  Polio Type 1 (antibody threshold ≥1:8) (n=61,64) | 100.00 [94.13 to 100.00] | 100.00 [94.40 to 100.00]
  Polio Type 2 (antibody threshold ≥1:8) (n=61,64) | 98.36 [91.20 to 99.96] | 100.00 [9.40 to 100.00]
  Polio Type 3 (antibody threshold ≥1:8) (n=61,63) | 98.36 [91.20 to 99.96] | 100.00 [94.31 to 100.00]
  Hepatitis b 10 mIU/mL (n=38,48) | 100.00 [90.75 to 100.00] | 100.00 [92.60 to 100.00]
  Pertussis - FHA 82.00 EU/MI (n=65,68) | 93.85 [84.99 to 98.30] | 95.59 [87.64 to 99.08]
  Pertussis - Pertussis Toxoid 43.00 EU/mL (n=65,68) | 89.23 [79.06 to 95.56] | 95.59 [87.64 to 99.08]
  Pertussis - Pertactin 18.00 EU/mL (n=65,68) | 96.92 [89.32 to 99.63] | 95.59 [87.64 to 99.08]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Haemophilus influenzae type b the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.15 µg/mL threshold was calculated; Test type: Superiority or Other; Difference = 3.08, 95% CI [-7.22 to 13.73]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Haemophilus influenzae type b the difference in percentage between the two groups (13vPnC - 7vPnC) at 1.0 µg/mL threshold was calculated; Test type: Superiority or Other; Difference = 7.02, 95% CI [-7.28 to 21.14]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Diphtheria the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.01 IU/mL and 0.1 IU/mL thresholds was calculated; Test type: Superiority or Other; Difference = 0.00, 95% CI [-9.38 to 7.73]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Tetanus the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.01 IU/mL and 0.1 IU/mL thresholds was calculated; Test type: Superiority or Other; Difference = 0.00, 95% CI [-9.38 to 7.73]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Polio Type 1 the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 threshold was calculated; Test type: Superiority or Other; Difference = 0.00, 95% CI [-5.97 to 5.68]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Polio Type 2 the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 threshold was calculated; Test type: Superiority or Other; Difference = -1.64, 95% CI [-8.80 to 4.24]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For Polio Type 3 the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 threshold was calculated; Test type: Superiority or Other; Difference = -1.64, 95% CI [-8.80 to 4.21]
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; For Hepatitis b the difference in percentage between the two groups (13vPnC - 7vPnC) at 10 mIU/mL threshold was calculated; Test type: Superiority or Other; Difference = 0.00, 95% CI [-9.38 to 7.73]
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; For Pertussis - FHA the difference in percentage between the two groups (13vPnC - 7vPnC) at 82.00 EU/MI threshold was calculated; Test type: Superiority or Other; Difference = -1.74, 95% CI [-11.00 to 6.99]
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; For Pertussis - PT the difference in percentage between the two groups (13vPnC - 7vPnC) at 43.00 EU/mL threshold was calculated; Test type: Superiority or Other; Difference = -6.36, 95% CI [-17.03 to 3.16]
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; For Pertussis - Pertactin the difference in percentage between the two groups (13vPnC - 7vPnC) at 18.00 EU/mL threshold was calculated; Test type: Superiority or Other; Difference = 1.33, 95% CI [-6.79 to 9.68]

8. Secondary Outcome: Geometric Mean Antibody Concentration of Haemophilus Influenzae Type b in 13vPnC Group Relative to 7vPnC Group After the Infant Series
Time Frame: one month after the infant series (7 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (N)= number of participants with a determinate antibody concentration for the specified concomitant vaccine component.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 84 | 87
μg/mL | 1.99 [1.34 to 2.97] | 1.64 [1.09 to 2.47]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Test type: Superiority or Other; Ratio = 1.21, 95% CI 2-sided [0.69 to 2.14]

9. Secondary Outcome: Geometric Mean Antibody Concentration of Hepatitis B in 13vPnC Group Relative to 7vPnC Group After the Infant Series
Description: GMCs of anti-hepatitis B surface antigen (HBsAg) using a Food and Drug Administration (FDA) approved in vitro diagnostic kit are presented.
Time Frame: one month after the infant series (7 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (N)=number of participants with a determinate antibody concentration for the specified concomitant vaccine component.
Measure: Geometric Mean (95% Confidence Interval); unit: milli International Units (mIU)/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 38 | 48
milli International Units (mIU)/mL | 1257.74 [904.77 to 1748.42] | 1300.01 [976.91 to 1729.99]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Test type: Superiority or Other; Ratio = 0.97, 95% CI 2-sided [0.63 to 1.48]

10. Secondary Outcome: Geometric Mean Antibody Concentration Diphtheria Toxoid and Anti-Tetanus Toxoid in 13vPnC Group Relative to 7vPnC Group After the Infant Series
Time Frame: one month after the infant series (7 months of age)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- 13vPnC: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 2, 4, 6 months (infant series).
- 7vPnC: Participants received one single 0.5mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with ActHIB and Pediarix at 2, 4, 6 months (infant series).
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 38 | 48
IU/mL
  Diphtheria Toxoid | 0.86 [0.65 to 1.14] | 1.04 [0.80 to 1.34]
  Anti-Tetanus Toxoid | 0.93 [0.72 to 1.22] | 0.97 [0.73 to 1.28]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Test type: Superiority or Other; Ratio = 0.83, 95% CI 2-sided [0.57 to 1.21]

11. Secondary Outcome: Geometric Mean Antibody Concentration of Polio in 13vPnC Group Relative to 7vPnC Group After the Infant Series
Time Frame: one month after the infant series (7 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n)= number of participants with a postinfant series blood sample.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 94 | 108
titer
  Polio Type 1 (n=61,64) | 483.72 [352.52 to 663.75] | 479.79 [361.79 to 636.26]
  Polio Type 2 (n=61,64) | 368.26 [250.75 to 540.84] | 403.45 [249.90 to 551.96]
  Polio Type 3 (n=61,63) | 914.01 [638.80 to 1307.80] | 812.75 [577.32 to 1144.18]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Polio Type 1; Test type: Superiority or Other; Ratio = 1.01, 95% CI 2-sided [0.66 to 1.53]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Polio Type 2; Test type: Superiority or Other; Ratio = 0.91, 95% CI 2-sided [0.56 to 1.49]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Polio Type 3; Test type: Superiority or Other; Ratio = 1.12, 95% CI 2-sided [0.69 to 1.84]

12. Secondary Outcome: Geometric Mean Antibody Concentration of Pertussis Antigens in 13vPnC Group Relative to 7vPnC Group After the Infant Series
Time Frame: one month after the infant series (7 months of age)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 65 | 68
EU/mL
  Pertussis - filamentous hemagglutinin (FHA) | 207.85 [178.72 to 241.74] | 225.12 [191.97 to 264.01]
  Pertussis - pertussis toxoid (PT) | 98.68 [82.89 to 117.49] | 96.58 [86.45 to 107.89]
  Pertussis - pertactin | 141.23 [113.02 to 176.48] | 135.51 [107.13 to 171.41]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Pertussis - FHA; Test type: Superiority or Other; Ratio = 0.92, 95% CI 2-sided [0.74 to 1.15]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Pertussis - PT; Test type: Superiority or Other; Ratio = 1.02, 95% CI 2-sided [0.83 to 1.25]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Pertussis - Pertactin; Test type: Superiority or Other; Ratio = 1.04, 95% CI 2-sided [0.76 to 1.44]

13. Secondary Outcome: Percentage of Participants Achieving Antibody Titer (OPA) ≥1:8 in 13vPnC Group Relative to 7vPnC Group After the 3-Dose Infant Series
Description: Percentage of participants achieving functional antibody titer ≥1:8 as measured by opsonophagocytic activity assay (OPA) along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: one month after the infant series (7 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations;(n)=number of participants with a determinate postinfant series antibody titer to the given serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 94 | 108
Percentage of participants
  Common Serotypes - Serotype 4 (n=30,33) | 96.67 [82.78 to 99.92] | 100.00 [89.42 to 100.00]
  Common Serotypes - Serotype 6B (n=27,30) | 92.59 [75.71 to 99.09] | 93.33 [77.93 to 99.18]
  Common Serotypes - Serotype 9V (n=27,27) | 100.00 [87.23 to 100.00] | 100.00 [87.23 to 100.00]
  Common Serotypes - Serotype 14 (n=27,30) | 100.00 [87.23 to 100.00] | 100.00 [88.43 to 100.00]
  Common Serotypes - Serotype 18C (n=27,30) | 100.00 [87.23 to 100.00] | 96.67 [82.78 to 99.92]
  Common Serotypes - Serotype 19F (n=25,25) | 84.00 [63.92 to 95.46] | 80.00 [59.30 to 93.17]
  Common Serotypes - Serotype 23F (n=27,26) | 92.59 [75.71 to 99.09] | 100.00 [86.77 to 100.00]
  Additional Serotypes - Serotype 1 (n=30,32) | 83.33 [65.28 to 94.36] | 6.25 [0.77 to 20.81]
  Additional Serotypes - Serotype 3 (n=25,29) | 80.00 [59.30 to 93.17] | 3.45 [0.09 to 17.76]
  Additional Serotypes - Serotype 5 (n=30,33) | 100.00 [88.43 to 100.00] | 6.06 [0.74 to 20.23]
  Additional Serotypes - Serotype 6A (n=25,29) | 96.00 [79.65 to 99.90] | 48.28 [29.45 to 67.47]
  Additional Serotypes - Serotype 7F (n=22,24) | 100.00 [84.56 to 100.00] | 20.83 [7.13 to 42.15]
  Additional Serotypes - Serotype 19A (n=22,24) | 77.27 [54.63 to 92.18] | 12.50 [2.66 to 32.36]

14. Secondary Outcome: Percentage of Participants Achieving Antibody Titer (OPA) ≥1:8 in 13vPnC Group Relative to 7vPnC Group After the Toddler Dose
Description: Percentage of participants achieving functional antibody titer ≥1:8 as measured by opsonophagocytic activity assay (OPA) along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) were assessed. Results are reported for the serotypes with a determinate antibody titer.
Time Frame: One month after the toddler dose (13 to 16 months of age)
Population: All-available (per protocol) population consisting of eligible participants who had at least 1 valid and determinate assay result related to the proposed analysis; (n)= number of participants with determinant posttoddler dose antibody titer to the given serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 85 | 102
Percentage of participants
  Additional Serotypes - Serotype 6A (n=73,70) | 100.00 [95.1 to 100.00] | 90.0 [80.5 to 95.9]
  Additional Serotypes - Serotype 19A (n=71,72) | 100.00 [94.9 to 100.00] | 51.4 [39.3 to 63.3]

15. Secondary Outcome: Geometric Mean Antibody Titer (OPA) in 13vPnC Group Relative to 7vPnC Group After the Toddler Dose
Description: Antibody functionality/geometric mean titer (GMT) as measured by opsonophagocytic activity assay (OPA) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) were assessed. Results are reported for the serotypes with a determinate antibody titer.
Time Frame: One month after the Toddler Dose (13 to 16 months of age)
Population: All-available (per protocol) population consisting of eligible participants who had at least 1 valid and determinate assay result related to the proposed analysis; (n)=number of participants with a determinant antibody titer for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 85 | 102
titer
  Additional Serotypes - Serotype 6A (n=73,70) | 2147.58 [1630.73 to 2828.23] | 599.90 [375.83 to 957.54]
  Additional Serotypes - Serotype 19A (n=71,72) | 802.24 [633.92 to 1015.24] | 36.62 [21.09 to 63.59]

ADVERSE EVENTS:
Groups:
- 13vPnC Infant Series: Participants received one single 0.5mL dose of 13vPnC coadministered with ActHIB and Pediarix at 2, 4, 6 months (infant series).
- 7vPnC Infant Series: Participants received one single 0.5mL dose of 7vPnC coadministered with ActHIB and Pediarix at 2, 4, 6 months (infant series).
- 13vPnC 6-Month Follow-up: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with Haemophilus b Conjugate Vaccine (ActHIB) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined (Pediarix) at 2, 4, 6 months (infant series). Participants received one single 0.5mL dose of 13vPnC coadministered with ActHIB at 12-15 months of age (toddler dose).
- 7vPnC 6-Month Follow-up: Participants received one single 0.5mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with ActHIB and Pediarix at 2, 4, 6 months (infant series). Participants received one single 0.5mL dose of 7vPnC coadministered with ActHIB at 12-15 months of age (toddler dose).
Arm/Group | 13vPnC Infant Series | 7vPnC Infant Series | 13vPnC Toddler Dose | 7vPnC Toddler Dose | 13vPnC 6-Month Follow-up | 7vPnC 6-Month Follow-up
Serious Adverse Events (participants affected / at risk) | 9/120 | 9/126 | 1/86 | 0/103 | 4/86 | 1/103
Other Adverse Events (participants affected / at risk) | 104/120 | 110/126 | 33/86 | 51/103 | 20/86 | 33/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Infant Series (N=120) | 7vPnC Infant Series (N=126) | 13vPnC Toddler Dose (N=86) | 7vPnC Toddler Dose (N=103) | 13vPnC 6-Month Follow-up (N=86) | 7vPnC 6-Month Follow-up (N=103)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Bilateral otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 3 | 3 | 0 | 0 | 1 | 0
Bronchiolitis RSV (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Chairi I malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Complex febrile seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0 | 0
Febrile illness (fever) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Febrile seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fever of unknown origin (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumococcal meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia right middle lobe (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
RSV positive bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Right upper and left lower lobe pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rotaviral diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sensory integration disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (hand) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Tethered cord syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral URI (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Infant Series (N=120) | 7vPnC Infant Series (N=126) | 13vPnC Toddler Dose (N=86) | 7vPnC Toddler Dose (N=103) | 13vPnC 6-Month Follow-up (N=86) | 7vPnC 6-Month Follow-up (N=103)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Plagiocephaly (Congenital, familial and genetic disorders) | 2 | 3 | 0 | 0 | 0 | 0
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 2 | 1 | 0 | 0 | 0 | 0
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Macrocephaly (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 13 | 16 | 0 | 1 | 0 | 4
Dacryostenosis acquired (Eye disorders) | 3 | 2 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 17 | 2 | 6 | 0 | 2
Vomiting (Gastrointestinal disorders) | 8 | 10 | 1 | 6 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 8 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 4 | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 4 | 2 | 0 | 1 | 0 | 0
Teething (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infantile spitting up (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mouth cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 10 | 12 | 1 | 2 | 1 | 3
Irritability (General disorders) | 3 | 6 | 0 | 0 | 0 | 0
Granuloma (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Allergy to chemicals (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 57 | 65 | 8 | 10 | 5 | 12
Otitis media (Infections and infestations) | 40 | 37 | 1 | 10 | 9 | 14
Bronchiolitis (Infections and infestations) | 13 | 13 | 0 | 1 | 0 | 2
Otitis media acute (Infections and infestations) | 7 | 16 | 1 | 2 | 2 | 2
Viral infection (Infections and infestations) | 9 | 12 | 1 | 3 | 1 | 2
Candida nappy rash (Infections and infestations) | 8 | 7 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 6 | 8 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 7 | 4 | 0 | 0 | 2 | 4
Oral candidiasis (Infections and infestations) | 8 | 2 | 0 | 0 | 2 | 0
Croup infectious (Infections and infestations) | 3 | 6 | 3 | 1 | 1 | 4
Nasopharyngitis (Infections and infestations) | 4 | 5 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 5 | 0 | 0 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 4 | 3 | 0 | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 3 | 4 | 1 | 1 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 5 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 4 | 1 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 2 | 3 | 0 | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 4 | 1 | 0 | 1 | 1 | 2
Viral rash (Infections and infestations) | 3 | 2 | 1 | 2 | 2 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0
Roseola (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 2
Acute tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Dacryocystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Eczema infected (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Erythema infectiosum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpangina (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 4 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 2 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 1 | 1 | 1 | 0 | 0 | 0
Cardiac murmur functional (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 2
Food intolerance (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypervitaminosis a (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 2 | 0 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Penile blister (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 16 | 1 | 1 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 17 | 1 | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 3 | 3 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 1 | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0 | 1 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 0
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Macleod's syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 7 | 10 | 1 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 10 | 6 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 7 | 1 | 3 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Corrective lens user (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 0
Exposure to communicable disease (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Scleral hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Tinea capitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Speech disorder developmental (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Penile adhesion (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Acne infantile (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thalassaemia alpha (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis orbital (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eye disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 41/119 | 54/124 | 19/85 | 30/101 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (any)=present at site of vaccination.
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 31/110 | 43/118 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (any)
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 26/107 | 30/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (any)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 10/119 | 7/124 | 2/85 | 4/101 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement.
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 2/110 | 10/118 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 5/107 | 7/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)
Induration (Any) (Skin and subcutaneous tissue disorders) | 26/119 | 24/124 | 16/85 | 17/100 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (any)=present at site of vaccination.
Induration (Any) (Skin and subcutaneous tissue disorders) | 18/110 | 23/118 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (any)
Induration (Any) (Skin and subcutaneous tissue disorders) | 18/107 | 22/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (any)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 24/119 | 22/123 | 16/85 | 17/100 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (mild)=0.5 centimeters (cm) to 2.0 cm.
Induration (Mild) (Skin and subcutaneous tissue disorders) | 18/110 | 20/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (mild)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 18/107 | 20/116 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (mild)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 4/119 | 3/123 | 2/85 | 3/100 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (moderate)=2.5 cm to 7.0 cm.
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 4/110 | 4/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (moderate)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 0/107 | 5/116 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (moderate)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/119 | 0/123 | 0/85 | 0/100 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (severe) >7.0 cm.
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/110 | 0/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (severe)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/107 | 0/116 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (severe)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 25/119 | 24/124 | 21/85 | 19/100 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (any)=present at site of vaccination.
Erythema (Any) (Skin and subcutaneous tissue disorders) | 18/111 | 21/118 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (any)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 19/107 | 23/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (any)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 24/119 | 24/124 | 21/85 | 16/99 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (mild)=0.5 cm to 2.0 cm.
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 15/110 | 20/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (mild)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 17/106 | 21/116 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (mild)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 3/119 | 0/124 | 3/85 | 5/99 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (moderate)=2.5 cm to 7.0 cm.
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 3/108 | 0/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (moderate)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 1/106 | 3/116 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (moderate)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/119 | 0/124 | 0/85 | 0/99 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (severe) >7.0 cm.
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/108 | 0/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (severe)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/106 | 0/116 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (severe)
Fever ≥38°C but≤39°C (General disorders) | 19/114 | 20/121 | 11/78 | 12/94 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever ≥38 degrees C but ≤39 degrees C
Fever ≥38°C but≤39°C (General disorders) | 22/102 | 28/114 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥38 degrees C but ≤39 degrees C
Fever ≥38°C but≤39°C (General disorders) | 20/100 | 23/113 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥38 degrees C but ≤39 degrees C
Fever >39°C but≤40°C (General disorders) | 3/113 | 1/121 | 2/77 | 0/94 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >39 degrees C but ≤40 degrees C
Fever >39°C but≤40°C (General disorders) | 4/102 | 4/113 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >39 degrees C but ≤40 degrees C
Fever >39°C but≤40°C (General disorders) | 2/101 | 1/113 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >39 degrees C but ≤40 degrees C
Fever >40°C (General disorders) | 0/113 | 0/121 | 0/76 | 0/94 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >40 degrees C
Fever >40°C (General disorders) | 0/102 | 0/113 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >40 degrees C
Fever >40°C (General disorders) | 0/100 | 0/113 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >40 degrees C
Decreased appetite (General disorders) | 36/118 | 39/124 | 19/85 | 22/101 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 25/110 | 27/118 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 29/107 | 36/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Decreased sleep (General disorders) | 22/118 | 22/124 | 11/84 | 15/101 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Irritability
Decreased sleep (General disorders) | 27/110 | 23/118 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Decreased sleep (General disorders) | 23/107 | 22/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 67/119 | 67/124 | 24 | 44/101 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 47/111 | 55/118 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 37/107 | 48/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Irritability (General disorders) | 79/118 | 88/124 | 33/85 | 48/101 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 69/110 | 67/118 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 55/107 | 63/117 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.